CLINICAL TRIAL: NCT02658916
Title: A Multicenter, Open-Label, Long-Term Treatment Study of Intravenously Administered BIIB092 in Patients With Progressive Supranuclear Palsy Who Participated in Study CN002003
Brief Title: Extension Study of BIIB092 in Participants With Progressive Supranuclear Palsy (PSP) Who Participated in CN002003
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: 251PP301(NCT03068468) primary endpoint was not met;further development of Gosuranemab BIIB092 in progressive supranuclear palsy will not be pursued.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 251PP201; CN002-004 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-01-13; First posted 2016-01-20 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Supranuclear Palsy, Progressive
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — gosuranemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Panel 1: BIIB092 (Experimental): BIIB092 administered by intravenous (IV) infusion, once every four weeks.
  Interventions: Drug: BIIB092
- Panel 2: BIIB092 (Experimental): BIIB092 administered by intravenous (IV) infusion, once every four weeks.
  Interventions: Drug: BIIB092
- Panel 3: BIIB092 (Experimental): BIIB092 administered by intravenous (IV) infusion, once every four weeks.
  Interventions: Drug: BIIB092
- Panel 4: BIIB092 (Expansion Panel) (Experimental): BIIB092 administered by intravenous (IV) infusion, once every four weeks.
  Interventions: Drug: BIIB092

INTERVENTIONS:
Drug: BIIB092 — Same dose as corresponding CN002003 study panel.
  Other Names: BMS-986168

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of multiple intravenous (IV) infusions of BIIB092 in participants with Progressive Supranuclear Palsy (PSP). The study will also assess the pharmacodynamic (PD) effects of BIIB092 on cerebrospinal fluid (CSF) N-terminal tau, pharmacokinetics (PK), and immunogenicity of BIIB092 in participants with PSP.

DETAILED DESCRIPTION:
This study, previously posted by Bristol-Myers Squibb, has transitioned to Biogen under a licensing agreement.

ELIGIBILITY:
Key Inclusion Criteria:

1. Completed treatment in Study CN002003.
2. A diagnosis of probable or possible PSP consistent with Study CN002003 criteria with no new medical information or diagnoses since enrollment into Study CN002003 that might confer doubt on the PSP diagnosis.
3. Able to tolerate Magnetic Resonance Imaging (MRI).
4. Able to perform all protocol-specified assessments and comply with the study visit schedule.
5. Have reliable caregiver to accompany patient to all study visits. Caregiver must be able to read, understand, and speak local language fluently to ensure comprehension of informed consent and informant-based assessments of patient. Caregiver must also have frequent contact with patient (at least 3 hours per week at one time or at different times) and be willing to monitor the patient's health and concomitant medications throughout the study.
6. Patient must reside outside a skilled nursing facility or dementia care facility at the time of enrollment
7. Women of childbearing potential (WOCBP) and sexually active fertile men with partners who are WOCBP must use highly effective birth control.

Key Exclusion Criteria:

1. Presence of an unstable, clinically significant medical condition other than PSP including, but not limited to: hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal, immunological, psychological or neurological disease or malignancy.
2. Contraindication to undergoing a lumbar puncture (LP).
3. Recent drug or alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders (4th Edition).
4. Treatment with any investigational drugs (including placebo) other than BIIB092 or placebo given in Study CN002003 or devices within 90 days prior to enrollment
5. Any vaccination within 30 days prior to study drug administration.
6. Contraindication to the MRI examination for any reason
7. Any other sound medical, psychiatric, and/or social reason as determined by the investigator
8. Known history of human immunodeficiency virus.
9. Evidence of organ dysfunction or significant deterioration from prior values in CN002003 beyond what is consistent with the target population or that would place the patient at increased risk or risk of early study discontinuation.
10. Inability to be venipunctured and/or tolerate venous access.
11. History of allergy, hypersensitivity, or serious adverse reaction to monoclonal antibodies or related compounds or allergy to any of the components of the study drug

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 41 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs), AEs Leading to Discontinuation, Deaths | Day 1 through study completion (approximately 1.5 years or later)
Percentage of Participants with Marked Abnormalities in Clinical Laboratory Tests, Vital sign Measurements, ECGs, and Physical and Neurological Examinations | Day 1 through study completion (approximately 1.5 years or later)

SECONDARY OUTCOMES:
Serum Trough Concentration (C-trough) of BIIB092 | Up to study completion (approximately 1.5 years or later)
End-of-Infusion Serum Concentration of BIIB092 | Day 1 through study completion (approximately 1.5 years or later)
Number of Participants with drug antibodies (anti-BIIB092) in Serum | Up to study completion (approximately 1.5 years or later)
Percent Change from Baseline in Cerebrospinal Fluid (CSF) Concentrations of unbound N-terminal Tau at Week 48 | Baseline, Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (13):
- United States (13):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California, San Francisco, Medical Center at Parnassus, San Francisco, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Inc., Boca Raton, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas